CLINICAL TRIAL: NCT04149769
Title: Mobility and Therapeutic Benefits Resulting From Exoskeleton Use in a Home and Community Setting (SC140121 Study 3)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Michael Goldfarb, Professor Of Physical Medicine, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SC140121 Study 3
Record Dates: First submitted 2019-10-08; First posted 2019-11-04 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Poorly-ambulatory subjects previously enrolled in Studies 1 and/or 2, and as such will have prior experience walking in the exoskeleton.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Interventional (Other): Walking in an exoskeleton within the home and community.
  Interventions: Device: Indego Exoskeleton

INTERVENTIONS:
Device: Indego Exoskeleton — Regular dosing of Indego Exoskeleton walking.

SUMMARY:
The proposed study is a pilot study intended to inform the hypothesis that regular walking in an exoskeleton within the home and community might offer health benefit, neurological recovery, and/or mobility benefit to the user. This exploratory pilot study is also intended to assess the level of compliance (i.e., exoskeleton use) among study participants by characterizing extent the device is used beyond the minimum required.

DETAILED DESCRIPTION:
Study 3 Outline Study 3 enrollment will be limited to 1 or 2 subjects at each site. Each subject will take home an exoskeleton for the 8-week duration of the treatment period. The subjects will be selected from the pool of poorly-ambulatory subjects previously enrolled in Studies 1 and/or 2, and as such will have prior experience walking in the exoskeleton. Note that study 3 will emply the exoskeleton as per existing FDA approval (510(k) number K171334); specifically, "to enable individuals with spinal cord injury at levels T3 to L5 to perform ambulatory functions [in the home and community] with supervision of a specially trained companion in accordance with the user assessment and training certification program." Use of the exoskeleton in the home and community (i.e., outside a clinical setting) is referred to as "personal use." So that this study complies with FDA approval for personal use, subjects selected for enrollment in Study 3, along with each subject's designated support person, will be trained and certified for personal use in accordance with the manufacturer's FDA-approved personal use training program.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Size and limb proportions capable of fitting in the exoskeletal device :
* Height between 1.55 m (5 ft, 1 in) and 1.92 m (6 ft, 3 in).
* Femur length between 37.5 cm (15 in) and 43.125 cm (17.25 in).
* Body mass no greater than 114 kg (250 lb).
* "Poorly ambulatory" individual, defined as a person with FIM Gait 2- 6, who may be able to walk short distances with or without braces or stability aid, or may be able to walk with assistance of one person, but whose primary means of mobility is a manual or power-operated wheelchair.
* Sufficient upper extremity strength and coordination to balance using appropriate stability aids, such as a rolling walker or forearm crutches, during exoskeleton walking.
* Neurological injury level (NLI) T3 to L5 (between and inclusive).
* Chronic SCI: at least 6 months post-injury, and preferably post-injury more than 1 year.
* Sufficient bone health for walking with full weight-bearing without undue risk of fracture, as determined by each subject's personal medical doctor, and approved by each site's medical supervisor.
* Passive range of motion (PROM) at shoulders, trunk, upper extremities and lower extremities within functional limits for safe gait and use of appropriate assistive device/stability aid.
* Skin intact where interfacing with robotic device.
* MAS for spasticity score 3 or less in lower extremities.
* Resting blood pressure and heart rate within established guidelines for locomotor training, specifically systolic 150 mmHg or less, diastolic 90 mmHg or less, heart rate 105 bpm or less.
* Ability to tolerate an upright standing position for 20 min, passive or active, without being lightheaded or having a headache.
* Availability and willingness of support person to be trained in accordance with the FDA training protocol for personal use of the exoskeleton, and who will assume responsibility for the support person role, which specifically includes providing ambulatory support during all exoskeletal walking.
* Access to a wireless internet connection (for use of exoskeleton iPod device).
* Willingness and ability to electronically send walking session reports from exoskeleton iPod to appointed site monitor following each walking session.

Exclusion Criteria:

* Heterotopic ossification that, in the opinion of the site medical supervisor, would place the subject at undue risk for fracture.
* Inability to follow instructions.
* Colostomy bag.
* Women who are pregnant or attempting to become pregnant during the course of the study. Note that a pregnancy test will be required and must be negative for all women prior to enrolling in the study, and will be additionally required and must be negative every four weeks during the course of the study protocol.
* Any disease, concomitant injury, or condition that interferes with the performance or interpretation of the protocol- specified assessments.
* Insufficient availability to complete study.
* Any other issue which, in the opinion of the investigators or medical supervisor, make the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Ten meter walk test (10MWT) | 18 weeks
  Measure of mobility (specifically gait speed) while wearing exoskeleton. Scale 1 to 7 (1=total assistance and 7=independent)
Six minute walk test (6MWT) | 18 weeks
  Measure of gait speed over six minutes while wearing exoskeleton. Scale 1 to 7 (1=total assistance and 7=independent)
Walking Index for Spinal Cord Injury II (WISCI-II) | 18 weeks
  Assessment of physical assistance required during walking while wearing exoskeleton. Scale 0 to 20 (0= unable to participate and 20 Ambulates with no devices, no braces and no physical assistance.
Functional Independence Measures (FIM) gait score | 18 weeks
  Assessment of physical assistance required during walking while wearing exoskeleton. Scale 0 to 7 (0= activity does not occur and 7= complete independence

SECONDARY OUTCOMES:
Timed Up and Go Test (TUG) | 18 weeks
  Measure of ability to stand, walk, turn, and sit while wearing exoskeleton. ≤ to 10 seconds to > 30 seconds (≤ 10 seconds=normal to > 30 predictive of requiring assistive device for ambulation and being dependent in ADLs
Borg Rating Scale of Perceived Exertion (RPE) | 18 weeks
  Measure of exertion required while using exoskeleton. Scale 6 to 20 (6= no exertion and 20 = maximal exertion
Modified Ashworth Score (MAS) | 18 weeks
  Measure of bone mineral density. Scale 0 to 4 (0=No increase in muscle tone and 4=Affected part(s) rigid in flexion or extension)
Bone Mineral Density | 18 weeks
  Measure of bone mineral density. Score -1 and above to -2.5 and below (-1.0 to +0.5= normal and -2.5 and below=osteoporosis)
Functional Reach | 18 weeks
  Measure of core strength. 0 to 3 (0= unable to reach 3=Reach > or = to 10 inches)
Manual Muscle Test (MMT) | 18 weeks
  Measure of muscle strength Scale 0 to 5 (0= No visible or palpable contraction and 5=Full ROM against gravity, maximul resistance
Ten Meter Walk Test without exoskeleton (10MWT) | 18 weeks
  Measure of walking speed without exoskeleton. Measure of mobility (specifically gait speed) while wearing exoskeleton. Scale 1 to 7 (1=total assistance and 7=independent)
Functional Independence Measures (FIM) gait score without exoskeleton | 18 weeks
  Measure of assistance required for walking without exoskeleton Scale 0 to 7 (0= activity does not occur and 7= complete independence
Walking Index for Spinal Cord Injury II (WISCI-II) score without exoskeleton | 18 weeks
  Measure of assistance required for walking without exoskeleton. Scale 0 to 20 (0= unable to participate and 20 Ambulates with no devices, no braces and no physical assistance.

OTHER OUTCOMES:
Spinal Cord Injury Spasticity Evaluation Tool (SCI-SET) | 18 weeks
  Survey of severity of spasticity. Score -3 to +3 ( -3 (extremely problematic) to +3 (extremely helpful).
Self-Report Survey | 18 weeks
  Survey of pain, spasticity, bowel and bladder function, and quality of life. Pain 0 to 5 (0=no pain and 5 =severe pain. Overall level of pain -3 to 3 (-3 =decreased and 3 =increased) Spasticity 0 to 5 (0= No spasticity and 5 Severe spasticity) Overall level of spasticity -3 to 3 (-3 =decreased and 3 =increased) Changes in bowel habits -3 to 3 (-3 worse and 3=better) Changes in bladder habits -3 to 3 (-3 worse and 3=better) Changes in mood -3 to 3 (-3 worse and 3=better)
American Spinal Injury Association (ASIA) Impairment Scale | 18 weeks
  Measure of neurological injury level and classification. Scale A to E (A= complete and E= normal)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldfarb, PhD, Principal Investigator — Vanderbilt University
Locations (3):
- United States (3):
  - Tampa VA, Tampa, Florida
  - Minnesota Mayo Clinic, Rochester, Minnesota
  - Vanderbilt University Medical Center, Nashville, Tennessee